CLINICAL TRIAL: NCT03869931
Title: Effects of Fenofibrate Administration in Patients With Diabetic Nephropathy
Brief Title: Effects of Fenofibrate Therapy in Diabetic Nephropathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGHDN001
Record Dates: First submitted 2019-02-28; First posted 2019-03-11 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus; Diabetic Nephropathies
Keywords: Fenofibrate; Diabetic Nephropathy; Metabolomics
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies | interventions — Fenofibrate

STUDY DESIGN:
Intervention Model Description: In this single-centre, open label study, 300 adults with DN will be recruited over 3 years. Following screening and baseline metabolic evaluations, eligible subjects will be treated with fenofibrate for 30-days and re-assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fenofibrate (Experimental): (Refer to intervention)
  Interventions: Drug: Fenofibrate

INTERVENTIONS:
Drug: Fenofibrate — Fenofibrate 100 mg or 300 mg (according to CrCl)

SUMMARY:
Diabetic nephropathy (DN) is a common cause of end-stage renal disease (ESRD) and accounts for nearly half of all new patients starting dialysis in Singapore, the country with the highest rates of DN in the Asia-Pacific region. Despite the scale of the problem, little progress has been made in our understanding of the pathogenesis of the disorder and no new therapies have been offered.

The investigators have conducted a metabolomics study of human diabetic nephropathy that revealed evidence for alterations in mitochondrial fuel metabolism in patients with the disease, a finding also reported in other recent studies of human DN. Based on this finding the investigators believe that dysregulated mitochondrial fuel oxidation is a major driver of diabetic nephropathy.

Fenofibrate is an agonist of peroxisome-proliferator activating receptor (ppar)-alpha that is approved for the treatment of hypercholesterolaemia and hypertriglyceridemia alone or combined in patients unresponsive to dietary and other non-drug therapeutic measures. Fenofibrate is also indicated for the reduction in the progression of diabetic retinopathy in patients with type 2 diabetes and existing diabetic retinopathy. Presently fenofibrate is not indicated for the treatment of diabetic nephropathy.

The investigators hypothesize that treatment with fenofibrate, taken orally at 300mg per day or 100mg per day for 30 days will lead to significant changes in the circulating metabolomics patterns in patients with DN. The investigators propose to administer the drug for a period of 30 days and will perform a comprehensive analysis of the state of fuel metabolism in these patients before, and after the administration of fenofibrate using targeted metabolomics and other approaches. Fundal photography, Optical Coherence Tomography (OCT) and Optical Coherence Tomography Angiography (OCTA) will also be performed at baseline and post-treatment. A total of 300 subjects will be recruited from Singapore General Hospital (SGH) Diabetes and Metabolic Centre. Our goal is to discover key changes in fuel metabolism in DN patients receiving fenofibrate.

DETAILED DESCRIPTION:
In this single-centre, open label study, 300 adults with DN will be recruited over 3 years. Following screening and baseline metabolic evaluations, eligible subjects will be treated with fenofibrate for 30-days and re-assessed.

4.1 Study Visits and Procedures Subjects will have their written informed consent taken during Visit 1 at the SGH Clinical Trials Research Centre (CTRC) and undergo screening and baseline assessments. Eligible subjects will return within the next 14 days for the initiation of study drug (Visit 2). The post-treatment and final visit (Visit 3) will take place 30 ± 7 days after Visit 2. Details of study visits are described in Table 1 (Refer study protocol).

4.1.1 VISIT 1: Informed Consent and Screening Interested patients will be scheduled for their first study visit (Visit 1) at SGH CTRC. Written informed consent will be taken by the principal or co-investigators assigned by the PI. After consent has been taken, study procedures in Table 1 will be performed. Subject will be given a sample copy of the treatment diary to familiarize them with the method to record study drug intake.

At the end of Visit 1, subjects will head over to Singapore Eye Research Institution (SERI) or Singapore National Eye Centre (SNEC)) for eye tests as mentioned in the following paragraphs.

Fundus Photography, conventional OCT and Assessment and grading of diabetic retinopathy (DR). The presence and severity of Diabetic Retinopathy (DR) or Diabetic Macular Edema (DME) will be assessed from digital fundus photographs and OCT. Following pupillary dilation, 7-field ETDRS photography using a non-mydriatic 45º fundus cameras will be obtained for each eye. The modified Wisconsin protocol will be used for DR grading. DR will be considered present if any characteristic lesion as defined by the ETDRS severity scale is present: microaneurysms (MA), hemorrhages, cotton wool spots, intraretinal microvascular abnormalities (IRMA), hard exudates (HE), venous beading, and new vessels. For each eye, a retinopathy severity score will be assigned according to a scale modified from the Airlie House classification system. Macular edema is defined by hard exudates in the presence of MA and blot hemorrhage within 1 disc diameter from the foveal center or presence of focal photocoagulation scars in the macular area. Clinically significant macular edema (CSME) is considered present when the macular edema involved is within 500 mm of the foveal center or if focal photocoagulation scars are present in the macular area. DR is categorized as minimal non-proliferative DR (level 20), mild non-proliferative DR (level 35), moderate non-proliferative DR (level 43 through 47), severe Non-proliferative Diabetic Retinopathy (NPDR) (level 53), and proliferative retinopathy (>60). Vision-threatening retinopathy is defined as the presence of severe NPDR, Proliferative Diabetic Retinopathy (PDR), or CSME. Presence of DME (centre involving and non centre involving) and central retinal thickness will also be assessed on OCT.

Ultrawide field (UWF) imaging Stereoscopic 200-degree-field ultrawide field images of each subject will be obtained using the Optos P200MA instrument. Unlike traditional fundus cameras, Optos imaging relies on proper eye positioning by the imager and correct patient fixation on a target, rather than the imager viewing the retinal structures for focus. The UWF200 images are centered on the fovea, covering approximately 25% and 82%, respectively, of the retinal area, including the optic disc, macula, and major vascular arcades. Grading of UWF imaging will be performed using the ETDRS protocol to determine the presence and severity of the following lesions: hemorrhages, microaneurysms, or both (H/Ma); intraretinal microvascular abnormalities (IRMA); venous beading (VB); cotton wool spots; hard exudates; retinal thickening; new vessels on the disc; new vessels elsewhere (NVE) on the retina; preretinal hemorrhage; vitreous hemorrhage; and traction retinal detachment. This test will be optional.

Optical Coherence Tomography (OCT) and Optical Coherence Tomography Angiography (OCTA) Spectral Domain Optical Coherence Tomography and optical coherence tomographic angiography will be performed in both eyes to obtain scans of the macular, macular thickness, retinal nerve fiber thickness optic disc, and optic nerve head.

4.1.2 Initiation of Study Drug

The PI or Co-Is assigned by the PI, will review screening results to determine whether subjects are eligible to continue with the study. Eligible subjects will be prescribed the study drug, fenofibrate (Trolip®). Fenofibrate is to be taken orally for 30 days, and the dose of fenofibrate will be adjusted based on the estimated CrCl during Visit 1 as below.

CrCl (ml/min) Fenofibrate Dosage > 60 300mg/day 30-59 100 mg/day < 30 Contraindicated

Study drug and subject treatment diary will be delivered to the subjects via a third party delivery service within 14 days from Visit 1. Alternatively, subjects can also return to the hospital to collect their study drug and drug diary. They will also be given a treatment diary to record the intake of study drug.

On the day of medication delivery or collection, the clinical research coordinator at SGH will call the subject to confirm that they have received the study drug. Subjects should not take the study drug until instructed by the clinical research coordinator. The clinical research coordinator will also check with subject if there is any change in their medication intake and is well feeling well before intake of the study drug.

They will be reminded to record intake of study drug into their treatment diary

4.1.3 VISIT 2: 4-Week Post-Treatment Visit

Visit 2 will take place 30 ± 7 days from the first dose of study drug. Subjects who are still on the study drug should continue take the study drug on the morning of Visit 2 with plain water. Subjects will be assessed to quantify changes in metabolic fuel utilization after treatment with fenofibrate. These changes are determined based on metabolomic profiling of acyl-carnitines, organic acids and amino acids and the eye tests.

SAMPLE COLLECTION

Up to a total of 47 ml (~3.2 tablespoons) of blood and 90 ml (~6.0 tablespoons) of urine will be collected for the entire study. During Visit 1 (Screening), approximately 25 ml (~1.7 tablespoons) of blood and 30 ml (~2.0 tablespoon) of urine will be collected. During Visit 2 (Dosing visit), 30 ml of urine will be collected and during Visit 3 (post-treatment & final visit), approximately 22ml (~1.5 tablespoon) of blood and 30 ml (~2.0 tablespoon) of urine will be collected.

Subjects who developed drug-related adverse reactions may require additional blood and urine taken for clinical assessment.

LABORATORY MEASUREMENTS

A) Blood Chemistry Screening and standard laboratory tests including full blood count, Potassium, Creatinine. alanine transaminase, aspartate transaminase, β-human chorionic gonadotropin, creatinine kinase (CK), lipid panel, glucose and HbA1c will be measured in the clinical laboratory using standard methods.

B) Metabolomic Profiling Metabolomic profiling of lipids, acylcarnitines (ACs), organic acids and ketones will be measured using liquid and gas chromatography and tandem mass spectrometry (LC-MS/MS and Gas Chromatography-MS/MS) at the Duke-National University of Singapore metabolomics laboratory.

ACs represent intermediaries of metabolic fuel oxidation and provides a "snap-shot" of in vivo metabolism at the cellular level. The measurement of the various long-, intermediate-chain ACs provide an indicator of fatty acid oxidation efficiency. Ceramides are toxic lipid intermediaries that are implicated in the pathogenesis of insulin resistance. Lactate, pyruvate, succinate, fumarate, malate, alpha-ketoglutarate and citrate are organic acids involved in tricarboxylic acid cycle activity. Beta hydroxybutyrate is a ketone which will also be measured with the organic acids.

C) Urine Protein Excretion

Urine ACR and PCR will be performed to quantify urine protein excretion.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 21 and 100 years of age
* Type 2 diabetes mellitus Increased urine protein excretion as defined as:
* More than one measurement in the past 1-year with urine microalbumin/creatinine ratio (ACR) > 3.3 mg/mmol creatinine, or urine total protein/creatinine ratio (PCR) > 0.2 g/urine creatinine, or creatinine clearance between 30-60 ml/min

More than one measurement in the past 1-year with urine microalbumin/creatinine ratio (ACR) > 3.3 mg/mmol creatinine or urine total protein/creatinine ratio (PCR) > 0.2 g/urine creatinine

* Known diabetes duration > 3 months
* HbA1c < 9%(within 3 months prior to enrolment)
* No change in dose of diabetes medications by more than two-fold or new agents added within the previous 3 months
* No change in dose of lipid-lowering medications by more than two-fold or new agents added within the previous 3 months
* Capable of providing informed consent

Exclusion Criteria

* Type 1 diabetes mellitus
* Known intolerance or allergic to statins
* Known intolerance or allergic to fenofibrate
* Known intolerance or allergic to peanut oil or soybean lecithin or related products
* Concurrent use of fibrates
* Concurrent use Colchicine
* Concurrent use Nicotinic Acid
* Concurrent use Cyclosporine
* Concurrent use Tacrolimus
* Concurrent use Amodiaquine
* Concurrent use Bile acid sequestrants
* Concurrent use Chenodiol
* Concurrent use Ciprofibrate
* Oral anticoagulants: vitamin K antagonist (e.g. warfarin), factor Xa inhibitors (eg. rivaroxaban, apixaban and dabigatran)
* Concurrent use Anti-obesity medications (e.g. phentermine, orlistat)
* Concurrent use Systemic steroids (e.g. prednisolone, hydrocortisone, dexamethasone)
* Hepatitis B
* Hepatitis C
* Autoimmune hepatitis
* Hemochromatosis
* Previous pancreatitis
* Serum alanine aminotransferase or aspartate aminotransferase above 2x upper limit of normal
* Serum creatinine kinase above upper limit of normal
* Creatinine clearance < 30 ml/min
* Renal replacement therapy
* Presence of any non-DN renal glomerular disease
* Any previous organ transplantation
* Previous bariatric surgery
* Gallbladder disease
* Untreated hypothyroidism
* Untreated thyrotoxicosis
* Hemoglobin < 10 g/L
* Any leukopenia
* Any thrombocytopenia)
* Cancer within the last 5 years (except basal cell carcinoma)
* Medical condition likely to limit survival to less than 3 years
* Currently participation in another clinical trial
* Pregnancy, or currently trying to become pregnant
* Nursing mothers
* Hospitalization within 1 month prior to enrolment
* Alcohol intake > 1 unit per day for women or > 2 units per day for men
* Any factors likely to limit adherence to interventions
* Any ongoing acute medical illness
* Failure to obtain informed consent from participant

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Serum concentration of palmitoylcarnitine following 30 days of fenofibrate treatment | Baseline and after 30 days of treatment
  Percentage change in serum concentration of palmitoylcarnitine following 30 days of fenofibrate treatment compared to baseline
Serum concentration of acetylcarnitine following 30 days of fenofibrate treatment | Baseline and after 30 days of treatment
  Percentage change in serum concentration of acetylcarnitine following 30 days of fenofibrate treatment compared to baseline
Serum concentration of leucine following 30 days of fenofibrate treatment | Baseline and after 30 days of treatment
  Percentage change in serum concentration of leucine following 30 days of fenofibrate treatment compared with baseline
Serum concentration of isoleucine following 30 days of fenofibrate treatment | Baseline and after 30 days of treatment
  Percentage change in serum concentration of isoleucine following 30 days of fenofibrate treatment compared with baseline
Serum concentration of valine following 30 days of fenofibrate treatment | Baseline and after 30 days of treatment
  Percentage change in serum concentration of valine following 30 days of fenofibrate treatment compared with baseline
Triglyceride concentration following 30 days of fenofibrate treatment | Baseline and after 30 days of treatment
  Absolute change in serum triglyceride (mmol/L) concentration following 30 days of fenofibrate treatment with baseline

SECONDARY OUTCOMES:
Change in ETDRS scale following 30 days of fenofibrate treatment | Baseline and after 30 days of treatment
  Change in ETDRS scale following 30 days of fenofibrate treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hong Chang Tan, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ansquer JC, Foucher C, Rattier S, Taskinen MR, Steiner G; DAIS Investigators. Fenofibrate reduces progression to microalbuminuria over 3 years in a placebo-controlled study in type 2 diabetes: results from the Diabetes Atherosclerosis Intervention Study (DAIS). Am J Kidney Dis. 2005 Mar;45(3):485-93. doi: 10.1053/j.ajkd.2004.11.004. PMID 15754270
- [Background] Keech A, Simes RJ, Barter P, Best J, Scott R, Taskinen MR, Forder P, Pillai A, Davis T, Glasziou P, Drury P, Kesaniemi YA, Sullivan D, Hunt D, Colman P, d'Emden M, Whiting M, Ehnholm C, Laakso M; FIELD study investigators. Effects of long-term fenofibrate therapy on cardiovascular events in 9795 people with type 2 diabetes mellitus (the FIELD study): randomised controlled trial. Lancet. 2005 Nov 26;366(9500):1849-61. doi: 10.1016/S0140-6736(05)67667-2. PMID 16310551
- [Background] Liu JJ, Ghosh S, Kovalik JP, Ching J, Choi HW, Tavintharan S, Ong CN, Sum CF, Summers SA, Tai ES, Lim SC. Profiling of Plasma Metabolites Suggests Altered Mitochondrial Fuel Usage and Remodeling of Sphingolipid Metabolism in Individuals With Type 2 Diabetes and Kidney Disease. Kidney Int Rep. 2016 Dec 16;2(3):470-480. doi: 10.1016/j.ekir.2016.12.003. eCollection 2017 May. PMID 29142974
- [Derived] Teo CHY, Lin MT, Lee IXY, Koh SK, Zhou L, Goh DS, Choi H, Koh HWL, Lam AYR, Lim PS, Mehta JS, Kovalik JP, Coffman TM, Tan HC, Liu YC. Oral Peroxisome Proliferator-Activated Receptor-alpha Agonist Enhances Corneal Nerve Regeneration in Patients With Type 2 Diabetes. Diabetes. 2023 Jul 1;72(7):932-946. doi: 10.2337/db22-0611. PMID 36445944